CLINICAL TRIAL: NCT01413126
Title: Acute and Second Meal Effects of Peanuts on Glycemic Response and Appetite in Obese Women With High Type 2 Diabetes Risk: a Randomized Crossover Trial
Brief Title: Peanuts Second Meal Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Rita de Cássia Gonçalves Alfenas, Federal University of Viçosa (Brazil)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NUTBRA
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Peanut; Blood glucose; Insulin; Non-esterified free fatty acids; Glucagon-like peptide-1; Peptide YY; Cholecystokinin; Appetitive; Food intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Peanut butter (Experimental): 42.5 g of Peanuts butter were added to a 75g available carbohydrate-matched breakfast meal
  Interventions: Dietary Supplement: Whole peanuts without skins, Peanut butter, or no peanuts (control)
- Whole peanut (Experimental): 42.5 g of whole peanuts were added to a 75g available carbohydrate-matched breakfast meal
  Interventions: Dietary Supplement: Whole peanuts without skins, Peanut butter, or no peanuts (control)
- No peanuts (control) (No Intervention)
  Interventions: Dietary Supplement: Whole peanuts without skins, Peanut butter, or no peanuts (control)

INTERVENTIONS:
Dietary Supplement: Whole peanuts without skins, Peanut butter, or no peanuts (control) — In accordance with the Food and Drug Administration qualified health claim regarding daily nut intake, 42.5 g of whole peanuts or peanut butter were added to a 75g available carbohydrate-matched breakfast meal each test session.

SUMMARY:
Nut consumption is associated with reduced risk of Type 2 diabetes. The aim of this study was to assess the effects of peanut (whole or peanut butter) to breakfast meals on glycemic, insulinemic and selected gut hormone responses, appetite, and food intake over two consecutive meals in obese women with high Type 2 diabetes risk. Fifteen women participated in a randomized crossover trial where 42.5g of whole peanuts (P), peanut butter (PB), or no peanuts (control-C) were added to a 75g available carbohydrate-matched breakfast meal. Postprandial concentrations of blood glucose, insulin, non-esterified free fatty acids (NEFA), glucagon-like peptide-1 (GLP-1), peptide YY (PYY), cholecystokinin (CCK), appetitive sensations and food intake were assessed after breakfast treatments and a standard lunch (75g available carbohydrate).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 30 - 35 kg/M2
* Not taking medications known to affect glycemia, fat metabolism, or appetite
* Regular breakfast consumer (≥100 kilocalories ingested within 2 hours of waking on ≥4d/wk)
* No body weight fluctuation (<5kg in the past 3 months)
* Willingness to eat all test foods
* No self-reported allergy to the foods provided in the study
* No self-reported sleep disorders
* At least one of the following conditions: waist circumference ≥ 88 cm; reported family history of Type 2 diabetes in first degree relatives; capillary glycemia between 5.5 - 7.0 mmol/L; and/or a 2-hour blood glucose of 7.8 - 11.1 mmol/L (impaired glucose tolerance)

Exclusion Criteria:

* Type 2 diabetes mellitus
* Dyslipidemia
* High blood pressure

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glucose homeostasis at eight hours | Baseline (-10), 15, 45, 60, 90, 120, 180, 240, 265, 295, 310, 340, 370, 430 and 490 minutes
  Postprandial concentrations and incremental area under the curve of blood glucose, insulin and glucagon-like peptide-1, and incremental area above the curve of non-esterified free fatty acids were assessed after breakfast treatments and a standard lunch

SECONDARY OUTCOMES:
Change from baseline in incretin hormones at four hours | Baseline (-10), 15, 45, 60, 90, 120, 180 and 240 minutes
  Postprandial concentrations and the incremental area under the curve of peptide YY and cholecystokinin were assessed after breakfast treatments
Change in food intake over 24 hours | 24 hours
  All food consumed in laboratory and after leaving the laboratory in the experiment day were recorded
Change from baseline in appetitive sensations at twelve hours | Baseline (-10), 15, 45, 60, 90, 120, 180, 240, 265, 295, 310, 340, 370, 430, 490, 550, 610, 670 and 730 minutes
  Appetite ratings were scored at baseline and in a pre-determined times on a 100 mm visual analogue scale anchored with descriptors of "not at all" and "extremely"

CONTACTS AND LOCATIONS:
Overall Officials: Caio EG Reis, PhD Student, Principal Investigator — University of Brasília, Brazil; Daniela N Ribeiro, M.Sc., Study Chair — Federal University of Viçosa, Brazil; Neuza MB Costa, Ph.D., Study Chair — Federal University of Espírito Santo, Brazil; Josefina Bressan, Ph.D., Study Chair — Federal University of Viçosa, Brazil; Rita CG Alfenas, Ph.D., Principal Investigator — Federal University of Viçosa, Brazil; Richard D Mattes, Ph.D., Study Director — Purdue University
Locations (1):
- Federal University of Viçosa, Viçosa, Minas Gerais, Brazil